CLINICAL TRIAL: NCT05750966
Title: Very Short-course Versus Standard Course Antibiotic Therapy in Patients With Acute ChOlangitis After Adequate Endoscopic BiliaRy drAinage
Brief Title: Short-course Antibiotics vs Standard Course Antibiotics in Patients With Cholangitis
Acronym: COBRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Rogier P. Voermans, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022.0292; 2022-002624-12 (EudraCT Number); NL80410.029.22 (Other: NL number CCMO)
Record Dates: First submitted 2023-02-03; First posted 2023-03-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cholangitis
Keywords: antibiotics; randomized controlled trial
MeSH Terms: conditions — Cholangitis | interventions — Gentamicins; Cefuroxime; Ceftriaxone; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: This study is designed as an open-label multicenter non-inferiority RCT. Patients will be randomly assigned to the intervention group (one day of ABT after ERCP) or the comparator group (4 to 7 days of ABT after ERCP).
Masking Description: Patients and investigators will know in which group they are assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very short-course antibiotics (Experimental): The antibiotic regimens will be according to the local hospital's antibiotic guideline for cholangitis (e.g. dosage form, dosage, frequency)and/or the national SWAB guideline in the Netherlands. In the experimental group, duration of ABT after adequate drainage will be 1 day. The duration will be 4 days and can be extended to 7 days in case of gram-negative bacteraemia, according to the national SWAB guideline regarding gram-negative sepsis.
  Interventions: Drug: cefrtriaxone, gentamicin, cefuroxim, ciprofloxin or other antibiotics according to local guideline (24 hours)
- Standard course antibiotics (Active Comparator): The antibiotic regimens will be according to the local hospital's antibiotic guideline for cholangitis, which are based on the previously mentioned national SWAB guideline. This means that the type of ABT, dosage and frequency will be comparable to the experimental group.
  In the comparator group treatment duration with ABT after ERCP will be according to the international well known and widely used TG18. The duration will be 4 days and can be extended to 7 days in case of gram-negative bacteraemia, according to the national SWAB guideline regarding gram-negative sepsis.
  Interventions: Drug: cefrtriaxone, gentamicin, cefuroxim, ciprofloxin or other antibiotics according to local guideline (4 to 7 days)

INTERVENTIONS:
Drug: cefrtriaxone, gentamicin, cefuroxim, ciprofloxin or other antibiotics according to local guideline (24 hours) — The duration of antibiotics is 24 hours after adequate biliary drainage. The choice of antibiotics will be according to local protocol and/or national Dutch SWAB guidelines. The most common antibiotics are described above, but this can differ based on allergies, local protocol or previous cultures. Drug classes may include: aminoglycosides, carbapenems, cefalosporins, fluorquinolones, sulfonamides, penicillines.
  Other Names: ceftriaxone; gentamicin; cefuroxim; ciprofloxacin
  Arms: Very short-course antibiotics
Drug: cefrtriaxone, gentamicin, cefuroxim, ciprofloxin or other antibiotics according to local guideline (4 to 7 days) — The duration of antibiotics is 4 to 7 days after adequate biliary drainage. The choice of antibiotics will be according to local protocol and/or national Dutch SWAB guidelines. The most common antibiotics are described above, but this can differ based on allergies, local protocol or previous cultures. Drug classes may include: aminoglycosides, carbapenems, cefalosporins, fluorquinolones, sulfonamides, penicillines.
  Other Names: ceftriaxone; gentamicin; cefuroxim; ciprofloxacin
  Arms: Standard course antibiotics

SUMMARY:
The goal of this multicentre randomized controlled trial is to investigate if a very short-course of antibiotics (1 day) for cholangitis after adequate drainage is non-inferior with respect to clinical cure in comparison with a standard course of antibiotics (4 to 7 days). Secondary objectives include:

* Will a one-day course of antibiotics for cholangitis after adequate drainage be non-inferior with respect to relapse of cholangitis and mortality in comparison with a standard course of antibiotics?
* Will a one-day course of antibiotics for cholangitis after adequate drainage result in less adverse drug events in comparison with a standard course of antibiotics?
* Will a one-day course of antibiotics for cholangitis after adequate drainage reduce length of hospital stay?
* Will a one-day course of antibiotics for cholangitis after adequate drainage improve quality of life?
* Will a one-day course of antibiotics for cholangitis after adequate drainage be cost-effective?

DETAILED DESCRIPTION:
Acute cholangitis is an infection of the biliary tract which is managed with biliary drainage and antibiotic therapy (ABT). Currently the international Tokyo Guidelines 2018 (TG18) recommend 4 to 7 days of ABT after source control. The national SWAB guideline of 2020 suggests a course of one to 3 days after biliary drainage. There are no randomized studies to guide the duration of ABT for acute cholangitis. Our recent retrospective study in the Netherlands showed that a short course of ABT seems safe and more evidence is available showing that other bacterial infections, including abdominal and bloodstream infections, can be treated with a short antibiotic course than previously assumed. Hence, the hypothesis is that a very short-course of ABT for acute cholangitis is non-inferior to a course of 4 to 7 days after adequate biliary drainage.

This study is designed as a multicenter non-inferiority randomized controlled trial. Patients will be randomly assigned to the intervention group (one day of antibiotic therapy after ERCP) or the comparator group (4 to 7 days of antibiotic therapy after ERCP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute cholangitis due to common bile duct stones, benign or malignant distal biliary obstruction or distal biliary stent dysfunction (only stents in situ for a minimum of 30 days)
* ERCP with adequate biliary drainage (all common bile duct stones are removed and/or there is adequate flow of clear bile with or without a biliary stent(s))
* Absence of fever (temperature <38.5°C) or a decrease of body temperature of at least 1°C has occurred within 24 hours after ERCP
* Age ≥ 18 years
* Written informed consent (IC)

Exclusion Criteria:

* Other aetiologies of acute cholangitis (e.g. primary sclerosing cholangitis, (sub)hilar and/or intrahepatic strictures or hilar stents)
* A recurrent cholangitis (within 3 months)
* Patients with surgically altered anatomy (leading to biliary-enteric anastomosis)
* Concomitant pancreatitis, according to International Association of Pancreatology/American Pancreatic Association guidelines.[18] Acute pancreatitis is diagnosed in case of fulfilment of 2 out of 3 of the following criteria:

  * Upper abdominal pain
  * Serum amylase or lipase >3x ULN
  * Signs of acute pancreatitis on imaging
* Concomitant cholecystitis, according to TG18 criteria.[19] Acute cholecystitis is suspected in case one item in A is met and one item in B and C.

A. Local signs of inflammation

* A1: Murphy's sign
* A2: Right upper quadrant mass/pain/tenderness B. Systemic signs of inflammation
* B1: Fever
* B2: Elevated C-reactive protein
* B3: Elevated WBC count C. Imaging findings characteristic of acute cholecystitis

  * Concomitant liver abscess
  * Another additional infectious diagnosis
  * Admission on an Intensive Care Unit (ICU) at time of randomisation
  * Use of maintenance antimicrobial therapy
  * Use of immunosuppressants
  * Neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
clinical cure rate by day 14 after ERCP without relapse by day 30 | 30 days
  Clinical cure is defined as the absence of both fever (>38°C) and/or shaking chills, and initial presenting symptoms. Relapse is defined as the initiation of new antibiotic therapy for recurrent cholangitis, subsequent infection in the hepatic-pancreatic-biliary region, or any other subsequent infection possibly related to the initial episode of cholangitis.

SECONDARY OUTCOMES:
All-cause 90-day mortality. | 90 days
  Mortality, which includes all causes.
Relapse of cholangitis within 90 days | 90 days
  Relapse is defined as the initiation of new antibiotic therapy for recurrent cholangitis, subsequent infection in the hepatic-pancreatic-biliary region, or any other subsequent infection possibly related to the initial episode of cholangitis.
Rate of any other subsequent infection requiring antibiotic therapy within 90 days. | 90 days
  Subsequent infections excluding recurrent cholangitis.
Rate of subsequent infections with MDR bacteria or Clostridioides difficile within 90 days. | 90 days
  Subsequent infections, in particular due to resistant bacteria.
Rate of other adverse drug events within 14 days | 14 days
  Includes: rash, diarrhoea (defined as ≥3 x loose stools per day), liver function abnormalities (defined as ≥5 x upper limit of normal (ULN) elevation in alanine aminotransferase (ALT) or ≥2 x ULN elevation in alkaline phosphatase (ALP) or ≥3 x ULN elevation in ALT and simultaneous elevation of total bilirubin concentration exceeding 2 x ULN (according to European association for the Study of the Liver Clinical Practice Guidelines: Drug-induced liver injury) AND without evidence of persistent obstruction on imaging OR elevation of liver enzymes after initial decrease. Lastly, other adverse drug events includes acute kidney injury, defined as increase in serum creatinine by ≥26.5 micromol/L within 48 hours or increase in serum creatinine to ≥1.5 times baseline (according to Kidney Disease: Improving Global Outcomes guidelines).
Length of intensive care and hospital stay for the initial episode of cholangitis. | 30 days
  Length of IC and hospital stay defined in days.
Quality of life and health utility. | 90 days
  This will be evaluated using the RAND-36 and EQ-5D-5L at day 7, day 30 and day 90.
  Scale title (RAND-36): Research and Devevelopment-36 Minimum raw score: 45 Maximum raw score : 198 Higher scores mean a better outcome.
  Scale title (EQ-5D-5L): European Quality of Life-5 Dimensions-5 Levels score Minimum score: 11111 Maximum score: 55555 Higher scores mean a worse outcome.
Societal costs and cost-effectiveness/-utility | 90 days
  The costs per cured patient without relapse and the costs per quality adjusted life year (QALY) Scale Title: Quality Adjusted Life Year. One quality-adjusted life year (QALY) is equal to 1 year of life in perfect health.QALYs are calculated by estimating the years of life remaining for a patient following a particular treatment or intervention and weighting each year with a quality-of-life score (on a 0 to 1 scale).
  Minimum score: 0 Maximum score: 1 Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (31):
- Netherlands (31):
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Rijnstate Ziekenhuis, Arnhem, Gelderland
  - Radboud umc, Nijmegen, Gelderland
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Maastricht UMC+, Maastricht, Limburg
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Elisabeth Tweesteden Ziekenhuis, Tilburg, North Brabant
  - Amstelland Ziekenhuis, Amstelveen, North Holland
  - Amsterdam UMC, Amsterdam, North Holland
  - OLVG, Amsterdam, North Holland
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Dijklander Ziekenhuis, Hoorn, North Holland
  - Zaans Medisch Centrum, Zaandam, North Holland
  - Deventer Ziekenhuis, Deventer, Overijssel
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Isala, Zwolle, Overijssel
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Groene Hart Ziekenhuis, Gouda, South Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Alrijne Ziekenhuis, Leiderdorp, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Haaglanden Medisch Centrum, The Hague, South Holland
  - Meander MC, Amersfoort, Utrecht
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
  - Universitair Medisch Centrum Groningen, Groningen
  - Martini Ziekenhuis, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miura F, Okamoto K, Takada T, Strasberg SM, Asbun HJ, Pitt HA, Gomi H, Solomkin JS, Schlossberg D, Han HS, Kim MH, Hwang TL, Chen MF, Huang WS, Kiriyama S, Itoi T, Garden OJ, Liau KH, Horiguchi A, Liu KH, Su CH, Gouma DJ, Belli G, Dervenis C, Jagannath P, Chan ACW, Lau WY, Endo I, Suzuki K, Yoon YS, de Santibanes E, Gimenez ME, Jonas E, Singh H, Honda G, Asai K, Mori Y, Wada K, Higuchi R, Watanabe M, Rikiyama T, Sata N, Kano N, Umezawa A, Mukai S, Tokumura H, Hata J, Kozaka K, Iwashita Y, Hibi T, Yokoe M, Kimura T, Kitano S, Inomata M, Hirata K, Sumiyama Y, Inui K, Yamamoto M. Tokyo Guidelines 2018: initial management of acute biliary infection and flowchart for acute cholangitis. J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):31-40. doi: 10.1002/jhbp.509. Epub 2018 Jan 8. PMID 28941329
- [Background] Sieswerda E, Bax HI, Hoogerwerf JJ, de Boer MGJ, Boermeester M, Bonten MJM, Dekker D, van Wijk RG, Juffermans NP, Kuindersma M, van der Linden PD, Melles DC, Pickkers P, Schouten JA, Rebel JR, van Zanten ARH, Prins JM, Wiersinga WJ. The 2021 Dutch Working Party on Antibiotic Policy (SWAB) guidelines for empirical antibacterial therapy of sepsis in adults. BMC Infect Dis. 2022 Aug 11;22(1):687. doi: 10.1186/s12879-022-07653-3. PMID 35953772
- [Background] Haal S, Wielenga MCB, Fockens P, Leseman CA, Ponsioen CY, van Soest EJ, van Wanrooij RLJ, Sieswerda E, Voermans RP. Antibiotic Therapy of 3 Days May Be Sufficient After Biliary Drainage for Acute Cholangitis: A Systematic Review. Dig Dis Sci. 2021 Dec;66(12):4128-4139. doi: 10.1007/s10620-020-06820-3. Epub 2021 Jan 19. PMID 33462749